CLINICAL TRIAL: NCT02775474
Title: Does Intraoperative Methadone Prevent Postoperative Pain in Bariatric Surgery?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Felipe Chiodini Machado, MD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 52792616.9.0000.0068
Record Dates: First submitted 2016-05-12; First posted 2016-05-17 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Pain, Postoperative; Chronic Pain
Keywords: Methadone; Pain, Postoperative; Chronic Pain; Bariatric Surgery
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone (Experimental): Methadone used as anesthesia opioid: induction with 0,15 mg / kg intravenous methadone. Boluses of 0,05 mg / kg intravenous methadone as needed intraoperatively
  Interventions: Drug: Use of Intraoperative Intravenous Methadone
- Fentanyl (Active Comparator): Fentanyl used as anesthesia opioid: induction with 6 mcg / kg intravenous fentanyl. Boluses of 2 mug / kg intravenous fentanyl as needed intraoperatively
  Interventions: Drug: Use of Intraoperative Intravenous Fentanyl

INTERVENTIONS:
Drug: Use of Intraoperative Intravenous Methadone — The intervention group will be given intravenous methadone at a fixed induction dose (0,15 mg / kg) and intraoperative boluses as judged necessary by the anesthesiologist
  Other Names: Methadone
  Arms: Methadone
Drug: Use of Intraoperative Intravenous Fentanyl — The active control group will be given intravenous fentanyl at a fixed induction dose (6 mg / kg) and intraoperative boluses as judged necessary by the anesthesiologist
  Other Names: Methadone
  Arms: Fentanyl

SUMMARY:
The recent increase in obesity has led to an increase in the need for bariatric surgery. In this group of patients the postoperative pain management is of vital importance. One strategy to improve postoperative analgesia is the use of intraoperative methadone, specially in those patients which regional anesthesia is not feasible. There is evidence that the use of intraoperative methadone can lead to a analgesia lasting 24 to 36 hours, while not associated with increased side effects when compared to other opioids with short or intermediate duration of action. In this study the investigators will evaluate the efficacy of intraoperative methadone in reducing postoperative pain and opioid consumption.

DETAILED DESCRIPTION:
Despite recent developments in postoperative pain control, many patients still suffer from moderate to severe pain after surgery. It is estimated that postoperative severe pain occurs in 20 to 40% of surgical procedures. With the recent increase in obesity incidence in the last years, the need for bariatric surgical intervention is greater. The management of postoperative pain in obese patients is particularly important, since this population have increased susceptibility to cardiovascular, pulmonary and thromboembolic perioperatively.

One of the strategies to improve pain management in the perioperative period is the intraoperative use of intravenous methadone, given its pharmacokinetic profile, specially in those patients in which regional anesthesia is contraindicated. Methadone is an opioid μ (MOR) receptor agonist, also a glutamate antagonist by blocking the N-methyl-D-aspartate (NMDA) receptor and a reuptake of serotonin and noradrenaline inhibitor. Intraoperative analgesia generated by administration of 20 to 30 mg methadone can last 24 to 36 hours. There is also evidence that methadone at 0.2 to 0.3 mg / kg is not associated with an increased incidence of side effects compared to other opioids with short or intermediate duration of action, such as fentanyl, sufentanyl and morphine.

The aim of this study is to evaluate the efficacy of intraoperative methadone in reducing postoperative pain and opioid consumption in patients undergoing open gastroplasty with or without associated Roux Y. Patients will undergo standardized general anesthesia, and the opioid used in anesthesia induction is methadone 0.15 mg / kg fentanyl or 6 mcg / kg bolus with additional if necessary. After extubation a intravenous morphine patient controlled analgesia device will be already available in the operating room. Groups will be compared regarding opioid consumption, pain scores, side effects, patient satisfaction and development of chronic postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Open bariatric surgery
* No contraindications for any drugs used during the trial
* Read, understood and signed the informed consent

Exclusion Criteria:

* Laparoscopic bariatric surgery
* Known allergy to any drugs used during the trial
* Cardiovascular disease
* Creatinine clearance lower than 60 mL/min/1.73 m2
* Chronic usage of opioids
* History of personality disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | Until 3 months postoperatively
  Postoperative pain will be evaluated using a verbal numerical pain scale (ranging from 0 to 10)

SECONDARY OUTCOMES:
Postoperative opioid consumption | Until 3 months postoperatively
  Postoperative opioid consumption will be evaluated at fixed postoperative times: 2h, 6h, 24h, 48h, 72h and 3 months
Side effects | Until 3 months postoperatively
  Nausea, vomiting, itching, urinary retention, respiratory depression, sedation will be evaluated at fixed postoperative times: 2h, 6h, 24h, 48h, 72h and 3 months
Chronic postoperative pain | 3 months postoperatively
  Patients will be evaluated for chronic pain 3 months postoperatively through a questionnaire which includes questions about numerical verbal scale of pain in the last three months, analgesic consumption and satisfaction with analgesia regimen

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Palmeira, MD, PhD, Study Chair — University of Sao Paulo General Hospital; Hazem Ashmawi, MD, PhD, Study Director — University of Sao Paulo General Hospital
Locations (1):
- Hospital das Clínicas da FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gourlay GK, Wilson PR, Glynn CJ. Methadone produces prolonged postoperative analgesia. Br Med J (Clin Res Ed). 1982 Feb 27;284(6316):630-1. doi: 10.1136/bmj.284.6316.630. No abstract available. PMID 6802264
- [Background] Shaiova L, Berger A, Blinderman CD, Bruera E, Davis MP, Derby S, Inturrisi C, Kalman J, Mehta D, Pappagallo M, Perlov E. Consensus guideline on parenteral methadone use in pain and palliative care. Palliat Support Care. 2008 Jun;6(2):165-76. doi: 10.1017/S1478951508000254. PMID 18501052
- [Background] Toombs JD, Kral LA. Methadone treatment for pain states. Am Fam Physician. 2005 Apr 1;71(7):1353-8. PMID 15832538
- [Background] Kharasch ED. Intraoperative methadone: rediscovery, reappraisal, and reinvigoration? Anesth Analg. 2011 Jan;112(1):13-6. doi: 10.1213/ANE.0b013e3181fec9a3. No abstract available. PMID 21173206
- [Background] Gourlay GK, Willis RJ, Wilson PR. Postoperative pain control with methadone: influence of supplementary methadone doses and blood concentration--response relationships. Anesthesiology. 1984 Jul;61(1):19-26. PMID 6742480
- [Background] Inturrisi CE. Pharmacology of methadone and its isomers. Minerva Anestesiol. 2005 Jul-Aug;71(7-8):435-7. PMID 16012416
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Udelsmann A, Maciel FG, Servian DC, Reis E, de Azevedo TM, Melo Mde S. Methadone and morphine during anesthesia induction for cardiac surgery. Repercussion in postoperative analgesia and prevalence of nausea and vomiting. Rev Bras Anestesiol. 2011 Nov-Dec;61(6):695-701. doi: 10.1016/S0034-7094(11)70078-2. English, Multiple languages. PMID 22063370
- [Background] Chui PT, Gin T. A double-blind randomised trial comparing postoperative analgesia after perioperative loading doses of methadone or morphine. Anaesth Intensive Care. 1992 Feb;20(1):46-51. doi: 10.1177/0310057X9202000109. PMID 1609941
- [Background] Richlin DM, Reuben SS. Postoperative pain control with methadone following lower abdominal surgery. J Clin Anesth. 1991 Mar-Apr;3(2):112-6. doi: 10.1016/0952-8180(91)90007-a. PMID 2039637
- [Result] Fernandez AZ Jr, Demaria EJ, Tichansky DS, Kellum JM, Wolfe LG, Meador J, Sugerman HJ. Multivariate analysis of risk factors for death following gastric bypass for treatment of morbid obesity. Ann Surg. 2004 May;239(5):698-702; discussion 702-3. doi: 10.1097/01.sla.0000124295.41578.ab. PMID 15082974